CLINICAL TRIAL: NCT06539429
Title: Phase I Clinical Study to Evaluate Safety and Efficacy of ANT-301 in Knee Osteoarthritis Patients
Brief Title: Clinical Study to Evaluate Efficacy and Safety of ANT-301 in Patients With Knee Osteoarthritis in Grade III/IV by K/L
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANT-301-102
Record Dates: First submitted 2024-04-30; First posted 2024-08-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ANT-301 (Experimental): Vial containing allogenic adipose-derived mesenchymal stem cells and human fibrin hydrogel
  Interventions: Biological: ANT-301

INTERVENTIONS:
Biological: ANT-301 — Administration on Day 1

SUMMARY:
This is a phase I open study to evaluate the efficacy and safety of ANT-301 in patients with knee osteoarthritis K&L Grade III/IV.

DETAILED DESCRIPTION:
Study Design: open-label, single-center, dose-escalation study

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been provided with information about the clinical trial and have provided written consent on the informed consent form
2. Patients aged 19 to 70 years old.
3. Patients diagnosed with K&L grade III/IV knee osteoarthritis
4. Patients with a VAS pain score of 40mm or higher when measured on a 100-point scale

Exclusion Criteria:

1. Patients with joint diseases other than osteoarthritis
2. Patients who have undergone knee joint surgery or radiation therapy to the knee joint within 6 months prior to the screening
3. Patients who received intra-articular injections within 6 months prior to the screening
4. Patients who have received systemic steroid therapy within 3 months prior to the screening
5. Patients who have received immunosuppressive agents within 3 months prior to the screening
6. Patients who have received cell therapy or gene therapy to the target knee within 5 years prior to the screening
7. Patients who are unwilling to use contraception during the clinical trial period

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Safety assessment | Week 2, 4, 8, 12, 24 and Month 12
  Number of Adverse events and Laboratory Abnormalities

SECONDARY OUTCOMES:
Pain improvement according to VAS scale measurements | Baseine, Week 4, 8, 12, 24 and Month 12
  The VAS scale ranges from 0 (no pain) to 10 (worst possible pain), with higher scores indicating worse pain.
IKDC score | Baseline, Week 4, 8, 12, 24 and 12 months
  IKDC subjective knee evaluation form scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
WOMAC questionnaire score | Baseline, Week 4, 8, 12, 24 and 12 months
  Difference in WOMAC questionnaire scores between baseline and each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No